CLINICAL TRIAL: NCT05187338
Title: Triplex CTLA4/PD1/PDL1 Checkpoint Inhibitors Combination Therapy for Advanced Solid Tumors
Brief Title: Triplex Checkpoint Inhibitors Therapy for Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZICI3-015
Record Dates: First submitted 2021-12-28; First posted 2022-01-11 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer; Liver Cancer; Colorectal Cancer; Pancreas Cancer; Ovary Cancer; Head and Neck Cancer; Breast Cancer; Gastric Cancer; Cervical Cancer; Esophageal Cancer; Sarcoma
Keywords: Solid tumor; CTLA4 antibody; PD1 antibody; PDL1 antibody; Interventional Radiology; Trans-artery infusion; Intra-tumor injection
MeSH Terms: conditions — Lung Neoplasms; Liver Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Head and Neck Neoplasms; Breast Neoplasms; Stomach Neoplasms; Uterine Cervical Neoplasms; Esophageal Neoplasms; Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 3 drugs (Experimental): Three antibodies combination against PD1, PDL1, and CTLA4.
  Interventions: Drug: ipilimumab +pembrolizumab +durvalumab

INTERVENTIONS:
Drug: ipilimumab +pembrolizumab +durvalumab — This study has 3 subgroups:
  1. Ipilimumab +pembrolizumab +durvalumab is administrated with a total dose of 1-2mg/kg via vein, every 3 weeks.
  2. Ipilimumab +pembrolizumab +durvalumab is administrated with a total dose of 1-2mg/kg via sustained (10min) micro-pump infusion via artery, every 3 weeks.
  3. Ipilimumab +pembrolizumab +durvalumab is administrated with a total dose of 50-150mg via intra-tumor fine needle injection in 5 min, every 3 weeks.

SUMMARY:
This trial is designed to investigate the safety, response rates and survival outcomes of patients with advanced solid tumors by infusion of CTLA4, PD1 and PDL1 antibodies combination through venous (IV), artery (IA) or intra-tumor (IT).

DETAILED DESCRIPTION:
Malignant solid tumors including lung and liver cancers are the most common malignancy worldwide, and their mortality rates are very high. China has a huge population base with about 4,000,000 new cancer cases each year. More than 60% of the solid tumors in China are diagnosed at mid-to-late stage and have lost the chance of surgery. Recently a lot of therapeutic strategies have been developed and applied to clinic including targeted therapy and immunotherapy, but the overall therapeutic efficiency is still low. It is very difficult to treat patients with recurrent/refractory/metastatic advanced solid cancers and more alternative therapies are urgently needed.

Antibodies against CTLA4, PD1 and PDL1 are representative drugs for the check-points inhibitory agents, and their clinical indications have been approved in various types of tumors, including advanced melanoma, non-small cell lung cancer, renal cell carcinoma, and classical Hodgkin's lymphoma and late recurrent head and neck squamous cell carcinoma patients, et al. Those drugs are regularly systemically administrated by vein infusion, however, local delivery of those drugs via interventional radiology technique including trans-artery or intra-tumor injection may increase the local drug concentration of the tumor, improve the efficacy, and reduce systemic adverse reactions. CTLA4 antibody ipilimumab has been widely effectively using to combine with PD1 or PDL1 antibody and this study is to combine ipilimumab, PD1 antibody and PDL1 antibody, so called triplex checkpoint inhibitors combination therapy, for advanced solid tumors. To the investigator's knowledge, no studies have been developed on the safety, efficacy and survival benefit of the triplex checkpoint inhibitors combination therapy for cancer patients. This phase I-II clinical trial is designed to assess the safety and survival benefit of ipilimumab, pembrolizumab and durvalumab combination on patients with advanced solid cancers, including PFS, ORR, DCR, and median survival time.

ELIGIBILITY:
Inclusion Criteria:

1. Cytohistological confirmation is required for diagnosis of cancer.
2. Signed informed consent before recruiting.
3. Age above 18 years with estimated survival over 3 months.
4. Child-Pugh class A or B/Child score > 7; ECOG score < 2
5. Tolerable coagulation function or reversible coagulation disorders
6. Laboratory examination test within 7 days prior to procedure: WBC≥3.0×10E9/L; Hb≥90g/L； PLT ≥50×10E9/L；INR < 2.3 or PT < 6 seconds above control；Cr ≤ 145.5 umul/L；Albumin > 28 g/L；Total bilirubin < 51 μmol/L
7. At least one tumor lesion meeting measurable disease criteria as determined by RECIST v1.1.
8. Birth control.
9. Willing and able to comply with scheduled visits, treatment plan and laboratory tests.

Exclusion Criteria:

1. Patients participated in clinical trials of equipment or drugs (signed informed consent) within 4 weeks;
2. Patients accompany by ascites, hepatic encephalopathy and esophageal and gastric varices bleeding;
3. Any serious accompanying disease, which is expected to have an unknown, impact on the prognosis, include heart disease, inadequately controlled diabetes and psychiatric disorders;
4. Patients accompanied with other tumors or past medical history of malignancy;
5. Pregnant or lactating patients, all patients participating in this trial must adopt appropriate birth control measures during treatment;
6. Patients have poor compliance.

   Any contraindications for hepatic arterial infusion procedure:

   A.Impaired clotting test (platelet count < 60000/mm3, prothrombin activity < 50%).

   B.Renal failure / insufficiency requiring hemo-or peritoneal dialysis. C.Known severe atheromatosis. D.Known uncontrolled blood hypertension (> 160/100 mm/Hg).
7. Allergic to contrast agent;
8. Any agents which could affect the absorption or pharmacokinetics of the study drugs
9. Other conditions that investigator decides not suitable for the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2029-10-30 (Estimated); Study Completion 2035-10-30 (Estimated)

PRIMARY OUTCOMES:
Safety of 3 drugs combination treatment | 5 years
  Safety will be assessed by recording all types of advise effects upon and after the treatment.
Progression-free survival | 5 years
  Progression-free survival (PFS) will be defined as the elapsed time from the first date of study treatment until documented disease progression (as per RECIST 1.1) or death from any cause, whichever is earlier. For patients who remain alive without progression, follow-up time will be censored at the date of last disease assessment.
Disease control rate | 5 years
  Disease control rate will be defined as objective response rate + steady disease rate.
Duration of remission (DOR) | 5 years
  DOR will be defined as the duration of the cancer remission.

SECONDARY OUTCOMES:
Overall survival | 5 years
  Overall survival (OS) will be defined as the elapsed time from the enrollment to death from any cause. For surviving patients, follow-up will be censored at the date of last contact (or last date known to be alive). Follow-up for OS will occur every 12 weeks (±1 month) until death or withdrawal of consent from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD, PHD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No